CLINICAL TRIAL: NCT00922324
Title: A Single-Center Randomized, Double-Blind, Placebo-Controlled Phase 1 Trial to Assess the Safety and Tolerability of Single and Multiple Daily Oral Administration of STP206 Live Biotherapeutic in Healthy Adult Subjects
Brief Title: Safety and Tolerability of STP206 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: STP206-001
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STP206 (Experimental): STP206 administered either as a single dose or as a daily dose for seven consecutive days
  Interventions: Drug: STP206 or vehicle control
- Vehicle Control (Placebo Comparator): STP206 vehicle administered as either a single dose or as a daily dose for 7 consecutive days
  Interventions: Drug: STP206 or vehicle control

INTERVENTIONS:
Drug: STP206 or vehicle control — STP206 or vehicle administered as either a single dose or as a daily dose for 7 consecutive days

SUMMARY:
The study will assess the safety, tolerability and fecal shedding of STP206 when given as a single dose and when given as daily doses for one week.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, 18 - 55 years of age
2. In general good heath as established by medical history, physical examination, and laboratory assessment
3. The subject is willing and able to comply with the protocol and complete all visits and procedures
4. Provide written informed consent after the nature of the study has been explained

Exclusion Criteria:

1. Subjects with any chronic illness or conditions that require treatment
2. Subjects with clinically significant abnormal laboratory values noted during the screening laboratory evaluation
3. Subjects with history of immune compromised conditions or any past use of immunosuppressant treatment
4. Subjects with current or past history of gastrointestinal disease, including any conditions with increased risk for bleeding (e.g., gingivitis, hemorrhoids)
5. Subjects who are lactose intolerant
6. Subjects who are intolerant or allergic to Splenda® or any of its ingredients (dextrose, maltodextrin, sucralose) or have a soy allergy
7. Subjects who have had a fever of 100°F or higher within the 2 weeks of the first dose of study drug
8. Subjects who have received a "live" vaccine within 30 days of the first dose of study drug
9. Subjects who have received any medications (prescription or OTC) within 2 weeks of the first dose of study drug
10. Subjects who have received and investigational drug with 30 days prior to the first dose of study drug
11. Subjects with a history of illicit drug use or alcohol abuse
12. Subjects with any other medical condition that may influence the objectives or outcomes of the study
13. Female subjects who are pregnant or lactating
14. Female subjects of childbearing potential who are not using an FDA approved birth control method
15. Subjects who are healthcare or daycare providers or those with close contact with immune compromised individuals
16. Subjects with a history of acute hepatitis, HIV infection or known to have positive diagnostic tests for HIV or HBV
17. Subjects who have a planned dental appointment from screening through 7 days after last dose of Investigational Product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | 7-days post dosing and 30-days post dosing
Changes in physical examination findings | 7-days post dosing
Changes in laboratory (hematology, chemistry, and urinalysis) variables | 7-days post dosing

SECONDARY OUTCOMES:
Fecal Shedding of STP206 components | 30 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Taha Keilani, MD, Study Director — Leadiant Biosciences, Inc.
Locations (1):
- SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States